CLINICAL TRIAL: NCT04424875
Title: Local Melatonin Application Following Removal of an Impacted Mandibular Third Molar: A Randomized Controlled Clinical Trial
Brief Title: The Effect of Melatonin Application Following Removal of Impacted Third Molar
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, lecturer,oral surgery, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Melatonin and 3rd molar
Record Dates: First submitted 2020-06-07; First posted 2020-06-11 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Impacted Third Molar Tooth
Keywords: impacted third molar; melatonine; bone healing
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study arm (Experimental): patients will undergo surgery to remove impacted lower third molar and receive Melatonin (3 mg melatonin into 2 ml hydroxyethyl cellulose gel 2%) in the socket following removal of the impacted third molar
  Interventions: Drug: 3 mg melatonin
- controlled arm (Placebo Comparator): patients will undergo surgery to remove impacted lower third molar and patients will receive no melatonin (2 ml of hydroxyethyl cellulose gel 2 %).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 3 mg melatonin — patients will remove impacted third molar and receive 3 mg melatonin into 2 ml hydroxyethyl cellulose gel 2%
  Other Names: melatonin group
  Arms: study arm
Drug: Placebo — patients will remove impacted third molar and receive 2 ml hydroxyethyl cellulose gel 2%
  Other Names: cellulose group
  Arms: controlled arm

SUMMARY:
In the present study, the main hypothesis hypothesizes that the local application of melatonin in the post-extraction socket produces favorable differences in the immediate postoperative period, as anti-inflammatory, analgesic, and early osteogenic regarding the natural healing process of the socket.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18ys
* no systemic disease
* impacted mandibular third molar class II position B on Pell- Gregory classification

Exclusion Criteria:

* history of metabolic or systemic diseases affecting bone or healing process,
* local infection,
* tobacco use,
* oral contraceptive,
* pregnancy and lactation
* patients who had taken analgesics or anti-inflammatories for 1 week prior to enrollment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Bone density | 6months
  The bone density within the extraction socket was measured using software of cone beam

SECONDARY OUTCOMES:
Osteoprotegerin (OPG) | 4weeks postoperatively
  Human Osteoprotegerin (OPG) ELISA Kit was used to detect OPG levels.The changes in OPG in the whole group in the predetermined period immediate postoperative , after 4 week,and 6months
pain sensation | 7 days postoperative
  a visual analogue scale (VAS) of 10 units in combination with a graphic rating scale. On the VAS, the left most end represented the absence of pain (score 0) and the right most end indicated the most severe pain (score 10).
swelling | 7 days postoperative
  a tape measure, from the tragus to the corner of the mouth.
trismus | 7days postoperative
  measuring the distance between incisal edges of upper and lower central incisor at maximal mouth

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cobo-Vazquez C, Fernandez-Tresguerres I, Ortega-Aranegui R, Lopez-Quiles J. Effects of local melatonin application on post-extraction sockets after third molar surgery. A pilot study. Med Oral Patol Oral Cir Bucal. 2014 Nov 1;19(6):e628-33. doi: 10.4317/medoral.19851. PMID 25350595